CLINICAL TRIAL: NCT01440127
Title: Randomized Clinical Trial Evaluating the Impact of Pretreatment With Metformin on Colorectal Cancer Stem Cells (CCSC) and Related Pharmacodynamic Markers
Brief Title: Impact of Pretreatment With Metformin on Colorectal Cancer Stem Cells (CCSC) and Related Pharmacodynamic Markers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to accrue all planned subjects in a timely fashion, but data collected will still be analyzed.
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Metformin CCSC
Record Dates: First submitted 2011-09-21; First posted 2011-09-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Subjects in this arm are randomized to receive metformin during the period of time between planning the surgery or biopsy and the actual procedure. After approximately 1 week of taking metformin, we will re-check the blood glucose. We will draw blood for cancer stem cells (about 2 teaspoons) and ask about symptoms. Subjects will stop taking metformin 2 days before the procedure.
  Interventions: Drug: Metformin
- Observation (No Intervention): No metformin will be given prior to the scheduled surgery or biopsy.

INTERVENTIONS:
Drug: Metformin — Pills will be taken for one week prior to the scheduled surgery or biopsy procedure.
  Other Names: Fortamet; Glucophage; Glumetza; Riomet
  Arms: Metformin

SUMMARY:
Metformin is drug that is normally used to treat people with diabetes. New research has discovered that metformin may also kill cancer stem cells. These cancer stem cells make up only a small portion of a cancer, but may be responsible for resistance to chemotherapy or for causing recurrence of the cancer. The purpose of this study is to determine the effect of metformin on colorectal cancer tumors. The study is designed to develop the methods to test tumors for cancer stem cells and then to determine the difference between treating with metformin and not treating with metformin with regard to the cancer stem cells. This research is investigational because the effect of metformin on cancer stem cells is not known in humans. Also, in patients who are not diabetic, metformin would normally not be given prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented colorectal cancer
* Intent to undergo disease resection or biopsy at least 7days from the treatment start date (allowing for a minimum of 5 days of treatment plus 2 days break)
* Medically fit for resection of their primary tumor or for biopsy
* Age 18-79 years
* Adequate renal function (serum creatinine levels <1.5 mg/dL [males], <1.4 mg/dL [females] or estimated creatinine clearance >= 60 ml/min)
* Adequate hepatic parameters, including aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 x upper limit of normal (ULN), total bilirubin ≤ 1.5 x ULN, and alkaline phosphatase levels ≤ 2.5 x ULN
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Intent to administer neoadjuvant chemotherapy or radiation therapy prior to the surgery or biopsy;
* Intent to perform surgery or biopsy within 7 days of study treatment start;
* Any situation where participation in this trial would alter, or cause significant risk of altering the ability or timing of a subject to undergo resection of their tumor
* Current use of metformin (within the past month);
* Blood glucose using point of care test < 70mg/dl;
* Renal disease or renal dysfunction not meeting inclusion criteria;
* Significant medical conditions such as cardiovascular collapse (shock), acute myocardial infarction, septicemia, acute or chronic metabolic acidosis
* History of, or states associated with, lactic acidosis such as shock or pulmonary insufficiency, alcoholism (acute or chronic), conditions associated with hypoxemia and pancreatitis
* Severe dehydration
* Clinical or laboratory evidence of hepatic disease
* Congestive heart failure requiring pharmacologic treatment, or unstable or acute congestive heart failure
* Known hypersensitivity to metformin hydrochloride
* Pregnant or lactating women
* Psychiatric illness or social situation that would limit compliance with study requirements and/or obscure results

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Expression of CD133 in tumors from patients treated or not treated with metformin | 2-weeks of metformin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wasif Saif, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States